CLINICAL TRIAL: NCT04821765
Title: A Phase II Study of PD-1 Antibody Combined With Chemoradiotherapy in Oligometastatic Esophageal Squamous Cell Carcinoma
Brief Title: Study of PD-1 Antibody Combined With Chemoradiotherapy in Oligometastatic Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XIN WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2749
Record Dates: First submitted 2021-03-15; First posted 2021-03-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Esophagus Cancer; Chemoradiotherapy; Oligometastatic Disease; Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — spartalizumab; Chemoradiotherapy; Albumin-Bound Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemoradiotherapy Combined With PD-1 Antibody (Experimental): The arm received chemoradiotherapy, 50-60Gy (BED) was given (1.8-2 Gy or 3-4Gy once daily , 5 days a week) to recurrent sites combined with chemotherapy（Cisplatin 75 mg/m2/day 1, and albumin paclitaxel 150 mg/m2/day 1 , every 3 weeks, 2 cycles ).PD-1 antibody (Tislelizumab) was performed simultaneously with concurrent chemoradiotherapy (Triprizumab 200mg，d1，every 3 weeks，2 cycles). After completion of chemoradiotherapy, PD-1 antibody was given continuously with 2-4 cycles of chemotherapy (the same regimen with concurrent chemotherapy) until 1 year or desease progression.
  Interventions: Drug: PD-1 antibody; Radiation: Chemoradiation; Drug: Albumin-Bound Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: PD-1 antibody — 200mg, d1, q3W
Radiation: Chemoradiation — 50-60Gy (BED) was given (1.8-2 Gy or 3-4Gy once daily , 5 days a week
Drug: Albumin-Bound Paclitaxel — 150mg/m2, d1, q3W
Drug: Cisplatin — 75mg/m2, d1, q3W

SUMMARY:
Chemoradiotherapy（CRT） is the main treatment for esophageal cancer patients with recurrent desease，and checkpoint blockade (PD-1) have been shown to be effective in advanced esophageal cancer. Therefore, PD-1 combined with chemoradiotherapy （CRT）may further improve the efficacy and become a new method for the treatment of esophageal cancer.This study intends to conduct a single-arm, prospective clinical study, aiming to evaluate the safety and efficacy of PD-1 combined with chemoradiotherapy(CRT) in patients with oligometastatic esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

•≥18 years；

* Esophageal squamous cell carcinomas；
* After radical treatment including surgery or definitive chemoradiotherapy
* Definition of oligometastases：≤3 metastases, including tumor beds and recurrent anastomotic sites；regional lymph node is defined as one metastatic site（AJCC8th, supraclavicular, mediastinal, abdominal）；metastases lesion in liver, lung, bone and brain is no more than 1.
* Karnofsky performance status(KPS)≥ 70；
* No immunotherapy were performed after recurrence；
* a white-cell count of at least 3500G/L, a hemoglobin concentration of at least 100 g/L, a platelet count of at least 100,000/lL, aspartate aminotransferase and alanine aminotransferase levels of within 1.5 times the upper limit of normal, a serum bilirubin level of 1.5 mg/dL or less, a creatinine level of 1.1 mg/dL or less;
* Hepatitis virus indicators: normal or hepatitis virus DNA titer less than 500 at the same time in an infectious disease hospital, and with the consent of the doctor can be treated；

Exclusion Criteria:

* Pregnancy, possible pregnancy, or breast-feeding;
* Psychological, family, social and other factors lead to uninformed consent;
* An esophageal mediastinal fistula and/or an esophageal tracheal fistula prior to treatment;
* Serious complications such as ischemic heart disease, arrhythmias, or other types of heart disease requiring treatment; liver cirrhosis; interstitial pneumonia or pulmonary fibrosis; active gastrointestinal bleeding; mental disorders being treated with antipsychoticagents or requiring treatment;
* Controlled diabetes mellitus;
* A history of autoimmune disease, autoimmune disease (such as colitis, hepatitis, hyperthyroidism, including but not limited to these disease or syndrome) and a history of immune deficiency, including test positive for HIV, or has other acquired, congenital immunodeficiency disease, or have a history of organ transplantation and the history of allogeneic bone marrow transplantation;
* A history of interstitial lung disease and a history of non-infectious pneumonia;
* Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 Copies /mL), hepatitis C ;(positive HCV antibody and HCV-RNA above the detection threshold of the assay）
* Any situation that is unstable or may compromise patient safety and compliance ;
* Active infections, such as active tuberculosis, are present;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Locoregional control rate | 3 year

SECONDARY OUTCOMES:
Number of participants with acute toxicities | 10 week, from the start of treatment to 1 month after chemoradiotherapy
  Acute toxicities are evaluated by NCI-CTC version 5.0
Tumor response rate | 2-3 months
Progression free survival | 1 year, 2 year, 3 year
Overall survival | 1 year, 2 year, 3 year
Objective response rate | 5.5 week
  Objective Response Rate are evaluated by RECIST 1.1
Radiomics analysis | 1 year, 2 year, 3 year, 5 year
  Analysis of correlation between radiomics signature extracted by LASSO and the rate of participants who achieve pathological complete response (pCR) and the overall survival based on MRI and CT simulation.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, Beijing Municipality
  - Department 4th of Radiation Oncology, Anyang Cancer Hospital, Anyang, Henan

IPD SHARING:
Plan to Share IPD: No